CLINICAL TRIAL: NCT03884218
Title: A Study to Assess Thermal Comfort of Frail Older People in a Care Home Setting.
Brief Title: Thermal Imaging in Old and Frail in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STH19634
Record Dates: First submitted 2019-03-13; First posted 2019-03-21 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Old Age; Debility
Keywords: Thermal Comfort
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal Comfort (Other): Infra red thermal image
  Interventions: Other: Infra red thermal imaging

INTERVENTIONS:
Other: Infra red thermal imaging — thermal image using a non-touch, non-ionising, thermal camera system

SUMMARY:
This study aims to test whether infrared thermal imaging using a non-touch, non-ionising, thermal camera system is feasible and reliable as an independent technique for thermal comfort assessment in older people and frail older people living in a care home and with or without mild cognitive impairment.

DETAILED DESCRIPTION:
Thermal comfort (TC) is a complex interaction involving physiological, social, cultural and clothing factors. In hospital and in care homes, health-issues (frailty, dementia, immobility) can affect a person's perception of TC.

In the UK 18,000 care homes provide living-communities for approximately 400,000 people. Many are old/frail and vulnerable to indoor chilling. A quality indicator for a good ''home'' environment is related to TC. However, in multiplyoccupied rooms TC varies between individuals. The challenge in health-assessment is in identifying ''uncomfortable'' residents (too hot/too cold). As TC is a subjective perception; a carer cannot reliably predict TC in another person.

The objectives are to use infra-red thermal imaging (IRTI) to 'see' the body temperature map, to demonstrate prevalence of TC/thermal discomfort, to demonstrate whether there is correspondence/dissociation between TC self-report and IRTI-measured body/extremity (hand) temperature.

The study aims to establish if TC can be predicted by an independent non-invasive imaging device

Expected achievements are a two-way pathway to health impact:

1. identification of eligible adults via NHS intermediary care- and awaiting care home residency
2. expert guidance and collaboration with NHS partners
3. translation of results from community to NHS setting e.g. stoke/aged care medicine for improved thermal care on the hospital wards Longer-term the expected achievement (5-7 years)-working with NHS colleagues and design/product development teams is expected to lead towards a commercialisation pathway.

ELIGIBILITY:
Inclusion Criteria:

Care home residents who are:

* Aged over 60 to a maximum age of 105 years
* Able to sit comfortably for up to 20 minutes without marked agitation.
* Ability to understand, read and speak English.

Exclusion Criteria:

Care home residents who are/have:

* Severe dementia
* Unable to hold a conversation
* Who do not wish to take part in the study
* Unable to speak or understand English
* Unable to sit with other residents
* Who are severely agitated or unsettled

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Thermometer | Baseline
  Body Temp: degrees
  whether an older persons perceptions about thermal comfort is best predicted by their body temperature from the thermometer in Degrees Centigrade. Their temp will be compared to their self reported thermal comfort.
Thermal Imaging comparison | Baseline
  whether an older persons perceptions about thermal comfort is best predicted by the image that the thermal camera provides (known as a thermal map) along with the data (temperature values) that can be extracted from the thermal image particularly over the area of interest which in this study is the hands and forearm. The thermal image will be compared to self-reported thermal comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Childs, Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided